CLINICAL TRIAL: NCT07084467
Title: Evaluation of First-Phase Ejection Fraction to Guide Cardiac Resynchronization Therapy - A Randomised Controlled Trial
Brief Title: A Study Testing a New Heart Scan Method to Improve Pacemaker Treatment for Heart Failure
Acronym: EFFECT-CRT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); King's College Hospital NHS Trust (Other); Barts Helth NHS Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25/LO/0562
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Resynchronisation Therapy (CRT); Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study will use single masking, meaning participants will not know whether they are in the EF1-guided or standard care group. The medical team adjusting the devices will know the group assignments because of the procedure involved. However, the investigators assessing echocardiograms and clinical results and outcomes will remain unaware (masked) of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care (SOC)
- EF1 optimisation (Experimental)
  Interventions: Other: EF1 guided CRT optimisation

INTERVENTIONS:
Other: EF1 guided CRT optimisation — In the EF1-guided optimisation group, the settings of the CRT device are adjusted to maximise early heart pumping efficiency, measured by a parameter called first-phase ejection fraction (EF1). Depending on the patient's heart rhythm, either the timing between heart chambers (AV or VV delay) is adjusted in small steps. The device setting that gives the best EF1 reading is chosen to help improve the heart's response to CRT.
  Arms: EF1 optimisation
Other: Standard of Care (SOC) — This group will receive standard of care for their health condition and CRT management.
  Arms: Standard of Care

SUMMARY:
Cardiac resynchronization therapy (CRT) is a device treatment for patients with heart failure which cannot be managed by medications alone. CRT can help the heart contract more efficiently and improve the pumping function. However, many patients do not benefit from this treatment. Therefore, a better selection tool will help us to determine the most suitable patients to receive this treatment. A new measure of pumping function of the heart called: first-phase ejection fraction or EF1 has been shown a good tool to select suitable patients for CRT. EF1 is a sensitive measurement of heart function and can be easily measured by echocardiography (an ultrasound heart scan).

The purpose of this study is to examine whether this new measurement (EF1) can predict outcomes and response to CRT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* On optimal medical therapy for heart failure
* Meets standard guideline criteria for CRT (including conduction system pacing), specifically:

  * NYHA class II to IV
  * Left ventricular ejection fraction (EF) ≤ 35%
  * QRS duration > 130 ms

Exclusion Criteria:

* Co-morbidities likely to reduce life expectancy to less than 6 months
* Major cardiovascular event within the past 6 weeks
* More than mild aortic stenosis
* Receiving continuous or intermittent infusion therapy for heart failure
* Poor ultrasound acoustic window preventing adequate imaging
* Unable to give informed consent
* Currently participating in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Volumetric response of left ventricle | 6 months post CRT implantation or 6 months post CRT optimisation
  This will be defined as a reduction in left ventricular end-systolic volume by more than 15% at following CRT implantation comparing to before CRT implantation on echocardiogram.

SECONDARY OUTCOMES:
Hospitalization for heart failure or all-cause death | From enrollment to 36 months post CRT implantation
  This composite endpoint will be collected over the entire duration of follow-up in the trial when the last patient randomized has reached 36 months of follow-up post CRT implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St. Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gu H, Li Y, Fok H, Simpson J, Kentish JC, Shah AM, Chowienczyk PJ. Reduced First-Phase Ejection Fraction and Sustained Myocardial Wall Stress in Hypertensive Patients With Diastolic Dysfunction: A Manifestation of Impaired Shortening Deactivation That Links Systolic to Diastolic Dysfunction and Preserves Systolic Ejection Fraction. Hypertension. 2017 Apr;69(4):633-640. doi: 10.1161/HYPERTENSIONAHA.116.08545. Epub 2017 Feb 21. PMID 28223475
- [Background] Gu H, Sidhu BS, Fang L, Webb J, Jackson T, Claridge S, Einarsen E, Razavi R, Papageorgiou N, Chow A, Bhattacharyya S, Chowienczyk P, Rinaldi CA. First-Phase Ejection Fraction Predicts Response to Cardiac Resynchronization Therapy and Adverse Outcomes. JACC Cardiovasc Imaging. 2021 Dec;14(12):2275-2285. doi: 10.1016/j.jcmg.2021.05.007. PMID 34886993
- [Background] Gu H, Cirillo C, Nabeebaccus AA, Sun Z, Fang L, Xie Y, Demir O, Desai N, He L, Lu Q, Nakou E, O'Gallagher K, Tountas C, Marvaki A, Monaghan M, Perera D, Pericao A, Ryan M, Sinclair H, Stylianidis V, Victor K, Wang B, Wang J, Wang R, Wu C, Yang Y, Yuan H, Zhang D, Zhang Y, Faconti L, Papachristidis A, Zhang L, Carr-White G, Shah AM, Xie M, Chowienczyk P. First-Phase Ejection Fraction, a Measure of Preclinical Heart Failure, Is Strongly Associated With Increased Mortality in Patients With COVID-19. Hypertension. 2021 Jun;77(6):2014-2022. doi: 10.1161/HYPERTENSIONAHA.121.17099. Epub 2021 May 10. PMID 33966447
- [Background] Bing R, Gu H, Chin C, Fang L, White A, Everett RJ, Spath NB, Park E, Jenkins WS, Shah AS, Mills NL, Flapan AD, Chambers JB, Newby DE, Chowienczyk P, Dweck MR. Determinants and prognostic value of echocardiographic first-phase ejection fraction in aortic stenosis. Heart. 2020 Aug;106(16):1236-1243. doi: 10.1136/heartjnl-2020-316684. Epub 2020 Apr 28. PMID 32345658
- [Background] Gu H, Saeed S, Boguslavskyi A, Carr-White G, Chambers JB, Chowienczyk P. First-Phase Ejection Fraction Is a Powerful Predictor of Adverse Events in Asymptomatic Patients With Aortic Stenosis and Preserved Total Ejection Fraction. JACC Cardiovasc Imaging. 2019 Jan;12(1):52-63. doi: 10.1016/j.jcmg.2018.08.037. Epub 2018 Nov 15. PMID 30448118
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. Circulation. 2017 Aug 8;136(6):e137-e161. doi: 10.1161/CIR.0000000000000509. Epub 2017 Apr 28. No abstract available. PMID 28455343